CLINICAL TRIAL: NCT01488123
Title: A Whole Systems Approach to the Study of Ayurveda for Cancer Survivorship, Project II
Brief Title: Integrative Approaches for Cancer Survivorship
Acronym: IACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: A112313; 5K23AT005340-03 (NIH)
Record Dates: First submitted 2011-12-05; First posted 2011-12-08 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Breast Cancer
Keywords: Breast, Cancer, Survivorship, Integrative, Complementary
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ayurvedic Intervention (Experimental)
  Interventions: Behavioral: Individualized manualized Ayurvedic intervention

INTERVENTIONS:
Behavioral: Individualized manualized Ayurvedic intervention — The manualized intervention will begin with an initial clinic visit (approximately 90 minutes) with the Ayurvedic practitioner in which the patient's diagnosis will be determined, an overview of Ayurveda will be given, and the initial treatment will be recommended based on the Ayurvedic diagnosis. Follow-up visits will range between 30 and 60 minutes in duration. The treatment modalities employed in the study will include nutrition, lifestyle, yoga, and marma (a treatment similar to acupressure).

SUMMARY:
The purpose of this study is to determine whether a four-month manualized Ayurvedic intervention will improve quality of life in recent breast cancer survivors.

DETAILED DESCRIPTION:
Cancer associated symptoms and impaired quality of life remain significant problems for patients despite advances in cancer treatment. Few effective treatment options exist for these symptoms. Integrative medicine is rising in popularity in the United States; however, few integrative medicine modalities have been rigorously studied. Ayurveda, a whole system of medicine that originated in the Indian subcontinent, has its own system of diagnostics and therapeutics, and among its strengths are wellness and prevention. We aim to perform a prospective single arm clinical study of a manualized Ayurvedic approach in breast cancer survivors with impaired quality of life. Specifically, we aim to develop the manualized Ayurvedic intervention; to assess feasibility; and to determine whether clinically meaningful effects can be achieved with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer survivor who is over 1 month and less than 12 months beyond the completion of primary therapy (surgery, radiation, and chemotherapy)
* Having received chemotherapy as part of their primary therapy for breast cancer
* Be in a complete remission
* Aged 18 years or older
* Able to read, write, and understand English
* Karnofsky Performance Status (KPS) 67 greater than 60.
* Ability to give informed consent

Exclusion Criteria:

* Having received Ayurvedic treatment within 2 months of study enrollment
* Receiving chemotherapy or radiotherapy at the time of study enrollment. Trastuzumab therapy is not exclusionary.
* Being within 1 month (before or after) of surgery for breast cancer (including breast reconstructive surgery). Smaller surgical procedures such as implant exchange are not exclusionary.
* Patients on adjuvant hormone therapy for less than 1 month

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-01; Primary Completion 2014-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in quality of life over 16 weeks | Baseline, End of week 8, End of week 16
  The investigators will use the EORTC QLQ C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire) 68 in conjunction with a breast cancer-specific subscale, BR23, to collect data on quality of life and cancer-related symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Anand Dhruva, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, Osher Center for Integrative Medicine, San Francisco, California, United States